CLINICAL TRIAL: NCT05427006
Title: Post Market Clinical Follow Up (PMCF) Medical Device Registry of Z-Systems Zirconia Dental Products: Z-Systems Registry Z-Systems Sub-Registry Plan: Z5-BL Dental Implants Z-Systems Sub-Registry Plan: Z5-TL Dental Implants
Brief Title: Post Market Clinical Follow Up (PMCF) Medical Device Registry of Z-Systems Zirconia Dental Products: Z-Systems Registry
Status: Recruiting | Type: Observational
Sponsor: Z-Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: Z-Systems Registry
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-05

CONDITIONS: Missing Teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Z5-BL Dental Implants
  Interventions: Device: Z5-BL Dental Implants
- Z5-TL Dental Implants
  Interventions: Device: Z5-TL Dental Implants

INTERVENTIONS:
Device: Z5-BL Dental Implants — This is an observational study, collecting data on the use of Z5-BL Dental Implants.
  Groups: Z5-BL Dental Implants
Device: Z5-TL Dental Implants — This is an observational study, collecting data on the use of Z5-BL Dental Implants.
  Groups: Z5-TL Dental Implants

SUMMARY:
Commercially pure (CP) titanium is the gold standard to produce dental implants because it has a huge volume of scientific publications over a period of more than 50 years, it is cheap and simple to produce (i.e., making dental implants economically "affordable") and comes in numerous specific designs of screws for various indications. That is why more than 95% of the implant market is dominated by titanium.

However, there is an innovation trend to manufacture implants from more inert and biocompatible materials. Ceramic implants represent a valuable alternative for expanding the patient base of clinicians, especially in cases with challenging aesthetic demand. Furthermore, there has been a significant increase in the number of patients requesting metal-free dentistry or bio-holistic implant treatments.

In the past, ceramics were often branded as "inferior" quality due to its reputation as being brittle but the growing volume of scientific publications specifically on zirconia are demonstrating that it is comparable in fracture-strength with titanium implants. There is a clear market niche for zirconia implants, especially in cases of:

* Aesthetic reconstructions in the anterior region, especially in patients with a thin gingival biotype
* Gingival recessions where a white colored implant is a great advantage
* For patients with a titanium intolerance/sensitivity
* For patients who prefer a bio-holistic/metal-free dental approach.

Today, clinicians are asking for long-term clinical results of zirconia as a dental implant material. Therefore, Z-Systems AG is conducting this zirconia dental implant registry. A registry design was chosen because it will capture long-term benefits/risks from clinical routine without patient selection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years) was or will be implanted with up to 5 implants of the Z-Systems Z5-BL or Z5-TLproduct group
* Patient has signed Informed Consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population are anyone needing to have their missing teeth replaced.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Absence of persistent subjective complaints | 12 months post-loading final prostheis
  Absence of persistent subjective complaints such as pain, foreign body sensation and/or dysesthesia
Absence of peri-implant infection | 12 months post-loading final prostheis
  Absence of peri-implant infection with suppuration
Absence of mobility | 12 months post-loading final prostheis
  Absence of mobility of dental implant

SECONDARY OUTCOMES:
Frequency of occurrence of device related Adverse Device Events (ADEs) and Serious Adverse Device Events (SADEs). | At implant surgery, 3 months, 6 months, 1-5 years post-loading with the final prosthesis (i.e., at every follow-up visit after implant surgery)
  Secondary Safety Outcome is frequency of occurrence of device related Adverse Device Events (ADEs), Serious Device Events (SADEs). Measured by asking patient if any adverse events occured since last follow-up.
Exploratory outcomes - complaints and incidence | At implant surgery, 3 months, 6 months, 1-5 years post-loading with the final prosthesis (i.e., at every follow-up visit after implant surgery)
  Rate of complaints and incidents related to the medical device during the whole registry.
Exploratory outcomes - clinical satisfaction | At implant surgery, 3 months, 6 months, 1-5 years post-loading with the final prosthesis (i.e., at every follow-up visit after implant surgery)
  Clinical satisfaction measured on a Likert scale: 1 to 6, with 1 being "not satisfied at all" to 6 being "highly satisfied.
Exploratory outcomes - patient satisfaction | At implant surgery, 3 months, 6 months, 1-5 years post-loading with the final prosthesis (i.e., at every follow-up visit after implant surgery)
  The patient's assessment of function and aesthetics is recorded by his/her assessment of function, aesthetic appearance, implants, speech and self-confidence. The parameters are assessed by rating the degree of satisfaction on a 100 mm Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Mariane Sordi, Study Director — Z-Systems
Locations (5):
- Germany (2):
  - MVZ Stiller GmbH, Berlin
  - Gemeinschaftspraxis Börner, Hagen, Köpenick
- Switzerland (3):
  - Praxis dentblanche AG, Solothurn, Grenchen
  - Praxis am Klosterplatz, Olten
  - HeilPraxis - ZahnMedizin, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Undecided